CLINICAL TRIAL: NCT07344363
Title: Prostate Cancer REsearch Using Cross-validation of Innovative Sampling, Integrating LC-MS/MS for Optimized Therapeutic Drug moNitoring
Acronym: PRECISION
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2025-012
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Applying Dried Blood Spots (DBS) techniques to pharmacokinetic analysis could significantly streamline the use of Therapeutic Drug Monitoring (TDM) in clinical practice. To establish DBS as a viable alternative sampling method, it is essential to demonstrate that results obtained from DBS analysis are reliable. This validation can be achieved through a cross-validation study. In this protocol, an original validated method, the plasma-based assay, serves as the "reference", while the alternative DBS-based analytical technique is the "comparator." The reliability will be defined analysing patients' samples with the new methods and comparing these results with those obtained with the reference LC-MS/MS (Liquid Chromatography-Mass Spectrometry) methods (in plasma). The possibility to apply DBS technique to pharmacokinetic analysis should largely facilitate the application of TDM to clinical practice.

DETAILED DESCRIPTION:
Applying Dried Blood Spots (DBS) techniques to pharmacokinetic analysis could significantly streamline the use of Therapeutic Drug Monitoring (TDM) in clinical practice. To establish DBS as a viable alternative sampling method, it is essential to demonstrate that results obtained from DBS analysis are reliable. This validation can be achieved through a cross-validation study. In this protocol, an original validated method, the plasma-based assay, serves as the "reference", while the alternative DBS-based analytical technique is the "comparator." The reliability will be defined analysing patients' samples with the new methods and comparing these results with those obtained with the reference LC-MS/MS methods (in plasma). The possibility to apply DBS technique to pharmacokinetic analysis should largely facilitate the application of TDM to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with abiraterone, apalutamide, darolutamide, and enzalutamide according to the dosing regimens described in the Summary of Product Characteristics. The treatment cycle does not matter but patients should be at the steady state (see section 4.2);• Age ≥18;
* Signed informed consent is required

Exclusion Criteria:

* Conditions that may limit the ability to adequately comply with the study procedures outlined in the protocol;
* Refusal of informed consent;
* Any condition that, in the investigator's judgment, could compromise appropriate participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with abiraterone, apalutamide, darolutamide, and enzalutamide according to the dosing regimens described in the Summary of Product Characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-11-19 (Estimated); Study Completion 2027-11-19 (Estimated)

PRIMARY OUTCOMES:
To assess the reliability of innovative analytical methods based on DBS sampling for the quantification of abiraterone, apalutamide, darolutamide, and enzalutamide | 24 months
  The reliability will be assessed comparing results obtained with the new methods and with the reference LC-MS/MS methods (in plasma) evaluating the comprehensive results of the following analysis:
  1. Calculation of Lin's concordance correlation coefficient (ρc) that quantifies the agreement between two measures of the same variable (e.g. chemical concentration);
  2. Quantification of the mean difference and of the limits of agreement between the two methods with Bland-Altman method;
  3. Evaluation of the slope and the intercept obtained using Passing-Bablok regression analysis;
  4. Check for agreement with FDA/EMA guidelines requirements: the difference between the results obtained with the new method and the results obtained with the gold standard assay (% difference) should be within 20% in least two-thirds (67%) of the samples analyzed

SECONDARY OUTCOMES:
To collect preliminary data regarding intra-patient (consecutive samples collected from the same patient) variability of Cmin values; | 24 months
  Intra-patient variation will be evaluated with intrapatient variation coefficient
To collect preliminary data regarding inter-patient (samples from different patients treated at the same drug dose) variability of Cmin values; | 24 months
  Inter-patient variation will be evaluated with variation coefficient
To conduct a preliminary evaluation of the correlation between drug exposure and toxicity | 24 months
  Mean difference in Cmin between patients with of without drug-related toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Riferimento Oncologico di Aviano (CRO), IRCCS, Aviano, Pordenone, Italy